CLINICAL TRIAL: NCT05871190
Title: The Effects Of Injectable Platelet-Rich Fibrin Application On Wound Healing Following Gingivectomy and Gingivoplasty Operations: Single-blind, Randomized Controlled, Prospective Clinical Study
Brief Title: The Effects Of I-PRF On Gingivectomy and Gingivoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Şeyma Çardakçı, Lecturer, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21.DUS.005
Record Dates: First submitted 2023-05-15; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Wound Heal
Keywords: VEGF, FGF-10, I-PRF,gingivectomy
MeSH Terms: interventions — proliferation regulatory factors, human urine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Active Comparator): I-PRF is placed on the wound site after a gingivectomy with the conventional method and closed with a periodontal dressing
  Interventions: Other: İnjectable platelet rich fibrin; Procedure: Gingivectomy anad gingivoplasty
- control group (Placebo Comparator): closure of the wound site with only a periodontal dressing after a gingivectomy with the conventional method.
  Interventions: Procedure: Gingivectomy anad gingivoplasty

INTERVENTIONS:
Other: İnjectable platelet rich fibrin — I-PRF is a type of platelet-rich fibrin (PRF) product obtained from the patient's own blood. PRF is a kind of tissue regeneration product of blood, rich in platelets, growth factors and cellular components.
  Other Names: i-prf
  Arms: Test group
Procedure: Gingivectomy anad gingivoplasty — leveling and regulation of the gingiva

SUMMARY:
The study aims to evaluate the effects of injectable platelet-rich fibrin (I-PRF) applications on early wound healing after gingivectomy and gingivoplasty surgery. In this randomized controlled single-blind study, gingivectomy and gingivoplasty surgeries were performed on 46 patients. The postoperative I-PRF-applied surgery areas were compared with control regions. The surgical areas were stained with Mira-2 tone and evaluated in the ImageJ program. Wound healing was evaluated by using the Modified Manchester Scar (MMS) scale and Landry, Turnbull, and Howley (LTH) index. Vascular endothelial growth factor (VEGF) and fibroblast growth factor 10 (FGF-10) concentrations were assessed by enzyme-linked immunoabsorbent assay (ELISA). The seven-day Visual Analog Scale was used to assess pain level.

Considering the results found, I-PRF applications revealed positive effects on epithelial wound healing after gingivectomy and gingivoplasty operations.

ELIGIBILITY:
Inclusion Criteria:

(a) systemically healthy patients ages 15-40 years, (b) pregnancy or lactation, (c) patients with chronic inflammatory gingival overgrowth in the mandibular and maxillary anterior area, (d) no attachment and bone loss, (e) not using immunosuppressive agents, systemic corticosteroids, chemotherapy, and/or radiotherapy drugs taken or prescribed 2 months before the study attempt, which may affect the study results, wound healing, and coagulation mechanism, and (f) patients with sufficient oral hygiene.

Exclusion Criteria:

(a) patients who had a history of periodontal treatment in the last 6 months, (b) smokers and alcohol users, those who used drugs that may cause gingival enlargement in the last 6 months, (c) patients with poor communication, and (d) patients who did not attend controls at designated times.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
effects of I-PRF on wound healing and epithelialization | seven months
  I-PRF applications revealed positive effects on epithelial wound healing after gingivectomy and gingivoplasty operations.

SECONDARY OUTCOMES:
effects of biochemical markers on wound healing | seven months
  In order to see the effects of biochemical markers on wound healing, gingival crevicular fluid samples should be taken at more frequent intervals.

CONTACTS AND LOCATIONS:
Overall Officials: şeyma ÇARDAKCI BAHAR, Lecturer, Principal Investigator — University of Health Sciences; Ankara, Turkey; Nebi Cansın KARAKAN, Asst. Prof., Study Director — Faculty of Dentistry Afyonkarahisar University of Health Sciences, Afyonkarahisar, Turkey; Ayhan VURMAZ, Assoc. Prof., Study Chair — Faculty of Medicine, Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey
Locations (1):
- University of Health Sciences; Ankara, Turkey, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year after the study was published